CLINICAL TRIAL: NCT04281875
Title: Assessing Benefits of Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Total Thyroidectomy.
Brief Title: Assessing Benefits of NIRAF Detection for Identifying Parathyroid Glands During Total Thyroidectomy.
Acronym: NIRAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carmen Solorzano, Professor of Surgery Chair, Department of Surgery Director, Vanderbilt Endocrine Surgery, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VICC HN 2017; 5R01CA212147-02 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Hypoparathyroidism; Thyroid Neoplasms; Thyroid Cancer
Keywords: Total Thyroidectomy; Intraoperative Parathyroid Identification; Near Infrared Autofluorescence; Postoperative Hypocalcemia; Postoperative Hypoparathyroidism
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: NIRAF detection technology is used as an adjunctive tool for intraoperative parathyroid identification in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND) in the interventional group.
  Generic Name of Device: Parathyroid Autofluorescence Detection Device (NIRAF detection technology).
  The Parathyroid Autofluorescence Detection Device consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nanometer (nm) laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 Milliwatts (mW). The device has an FDA clearance for clinical use in general surgeries and dermatological use (Class 2 device).
Who Masked: Participant
Masking Description: Only participants will be masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIRAF Detection Technology + (Experimental): Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).
  Interventions: Device: NIRAF Detection Technology
- NIRAF Detection Technology - (No Intervention): Parathyroid gland identification will be performed with the naked eye of the surgeon without using PTeye - NIRAF detection technology in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).

INTERVENTIONS:
Device: NIRAF Detection Technology — Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
  Other Names: PTeye Device
  Arms: NIRAF Detection Technology +

SUMMARY:
This study describes a single center, randomized, single-blinded clinical trial to assess the clinical benefits of the use of near infrared autofluorescence (NIRAF) detection with an FDA-cleared device 'Parathyroid Eye (PTeye)' for identifying parathyroid glands (PGs) during total thyroidectomy (TTx). It compares risk-benefits and outcomes in TTx patients where NIRAF detection with PTeye for parathyroid identification is either used or not used.

DETAILED DESCRIPTION:
Inadvertent damage or excision of a healthy parathyroid gland (PG) following a total thyroidectomy (TTx) could result in transient hypocalcemia (< 6 months) in 5 - 35% of cases or permanent hypocalcemia (> 6 months) in 7% of the patients (1, 2). In both of these circumstances, patients would require calcium and active vitamin D supplementation in addition to a potentially prolonged hospital stay and/or unplanned hospital readmission adding to unnecessary burden and healthcare costs. These complications could be minimized with label-free intraoperative PG identification using near infrared autofluorescence (NIRAF) detection with a fiber-probe based approach (3 - 5) as utilized in 'PTeye', which is medical device that was recently FDA-cleared (6). However, the true impact of this particular NIRAF-based approach on patient outcomes is yet to be determined

The aim of this prospective single blinded randomized study is to compare 2 groups of patients: TTx patients operated using NIRAF detection technology with PTeye as adjunct tool (NIRAF+) vs. patients operated without the adjunct technology (NIRAF-). The main objective of this study is to assess the benefit of intraoperative use of NIRAF detection technology via PTeye during TTx procedures with regard to postoperative hypocalcemia, PG identification, PG auto-transplantation and inadvertent resection rates compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

(i) All patients eligible for total thyroidectomy (TTx), with or without lymph node dissection. (includes patients undergoing a TTx who have undergone a prior neck exploration for parathyroid disease or other but have an intact thyroid).

(ii) All patients undergoing completion thyroidectomy.

Exclusion Criteria:

(i) Patients with concurrent parathyroid disease. (ii) Patients with incidental enlarged parathyroid discovered during TTx. (iii) Patients undergoing thyroid lobectomy/partial thyroidectomy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen C Solorzano, MD, FACS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Informed Consent Form and Clinical Study Report will be made available to other researchers as per the specified time-frame.
Supporting Information: ICF, CSR
Time Frame: Clinical Study Report will be shared 6 months after publication of trial data and will be available till end date of trial. Informed Consent Form will be shared for a year after the primary completion date of the trial.
Access Criteria: Request for Individual Patient Data (IPD) - Informed consent Form and Clinical Study Report - will be reviewed by the principal investigator of this clinical trial, before granting access to IPD

REFERENCES:
- [Background] Antakia R, Edafe O, Uttley L, Balasubramanian SP. Effectiveness of preventative and other surgical measures on hypocalcemia following bilateral thyroid surgery: a systematic review and meta-analysis. Thyroid. 2015 Jan;25(1):95-106. doi: 10.1089/thy.2014.0101. PMID 25203484
- [Background] Edafe O, Antakia R, Laskar N, Uttley L, Balasubramanian SP. Systematic review and meta-analysis of predictors of post-thyroidectomy hypocalcaemia. Br J Surg. 2014 Mar;101(4):307-20. doi: 10.1002/bjs.9384. Epub 2014 Jan 9. PMID 24402815
- [Background] McWade MA, Sanders ME, Broome JT, Solorzano CC, Mahadevan-Jansen A. Establishing the clinical utility of autofluorescence spectroscopy for parathyroid detection. Surgery. 2016 Jan;159(1):193-202. doi: 10.1016/j.surg.2015.06.047. Epub 2015 Oct 9. PMID 26454675
- [Background] Thomas G, McWade MA, Paras C, Mannoh EA, Sanders ME, White LM, Broome JT, Phay JE, Baregamian N, Solorzano CC, Mahadevan-Jansen A. Developing a Clinical Prototype to Guide Surgeons for Intraoperative Label-Free Identification of Parathyroid Glands in Real Time. Thyroid. 2018 Nov;28(11):1517-1531. doi: 10.1089/thy.2017.0716. Epub 2018 Sep 11. PMID 30084742
- [Background] Thomas G, McWade MA, Nguyen JQ, Sanders ME, Broome JT, Baregamian N, Solorzano CC, Mahadevan-Jansen A. Innovative surgical guidance for label-free real-time parathyroid identification. Surgery. 2019 Jan;165(1):114-123. doi: 10.1016/j.surg.2018.04.079. Epub 2018 Nov 12. PMID 30442424
- [Background] Voelker R. Devices Help Surgeons See Parathyroid Tissue. JAMA. 2018 Dec 4;320(21):2193. doi: 10.1001/jama.2018.18768. No abstract available. PMID 30512085
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Groups:
- NIRAF Detection Technology +: Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).
  NIRAF Detection Technology: Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
Period: Overall Study
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology - | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (14.1) | 46.4 (14.5) | 47.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 61 | 124
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 79 | 78 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 62 | 127
  Black | 13 | 17 | 30
  Asian | 1 | 0 | 1
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.9 (8.8) | 32.3 (8.4) | 32.1 (8.6)
Diagnosis [Count of Participants; unit: Participants]
  Graves' Diseases | 25 | 25 | 50
  Goiters and Nodular Diseases | 35 | 31 | 66
  Thyroid Cancers | 20 | 24 | 44
Preoperative calcium (pg/dL) [Mean (Standard Deviation); unit: pg/dL] | 9.5 (0.5) | 9.4 (0.4) | 9.5 (0.5)
Preoperative PTH (pg/mL) [Mean (Standard Deviation); unit: pg/mL] | 62.6 (28) | 81.1 (51.1) | 71.3 (40)
Preoperative vitamin D (mcg) [Mean (Standard Deviation); unit: mcg] | 29.5 (13) | 34.6 (20.6) | 32 (17.1)
Procedure [Count of Participants; unit: Participants]
  Total Thyroidectomy | 68 | 65 | 133
  Total Thyroidectomy with Central Neck Dissection | 8 | 12 | 20
  Reoperation | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Parathyroid Glands Identified With High Confidence Per Patient
Description: Average number of parathyroid glands identified (Experimental Group: Glands identified with naked eye + NIRAF; Control Group: Glands identified with naked eye) per patient
Time Frame: Immediate. During total thyroidectomy procedure.
Measure: Mean (Standard Deviation); unit: parathyroid glands
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
parathyroid glands | 2.81 (1.03) | 2.75 (0.95)
Statistical Analysis 1: Comparison: NIRAF Detection Technology + vs NIRAF Detection Technology -; Test type: Superiority; p = 0.6905, t-test, 2 sided

2. Secondary Outcome: Postoperative Hypoparathyroidism/Hypocalcemia (Permanent)
Description: If blood calcium has not normalized at 1st postsurgical clinical visit, total calcium level and/or PTH is subsequently measured as necessary. Patient is defined to have permanent hypoparathyroidism if PTH < 16 pg/mL and/or activated Vitamin D is required to be symptom free at or after the 6th postoperative month.
Time Frame: 6 months after total thyroidectomy
Population: Only participants with at least 6-months of follow-up were included in this analysis. The majority of follow-ups for thyroid surgery occured nat 5-14 days post-operation and most people do not return for longer follow-up unless they have on-going abnormal labs after that mark.
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

3. Secondary Outcome: Postoperative Hypoparathyroidism/Hypocalcemia (Transient)
Description: Undetectable postoperative PTH and/or low calcium (total calcium < 2mmol/L or 8 mg/dL, serum intact PTH < 16 pg/mL or 1 pmol/L) at first postoperative visit (usually 5-30 days after total thyroidectomy).
Time Frame: 5 days to 6 months after total thyroidectomy.
Population: Not all of the patients come back for follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 56 | 50
Participants | 3 | 5

4. Secondary Outcome: Postoperative Hypoparathyroidism/Hypocalcemia (Immediate)
Description: Postoperative low calcium (total calcium <8mg/dL or <2mmol/L) and/or undetectable parathyroid hormone (PTH) (serum intact PTH < 16 pg/mL or 1 pmol/L) within 24 hours after surgery
Time Frame: Within 24 hours after total thyroidectomy.
Population: 1 participant did not have their labs completed until 5-14 days post-operation.
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 79
Participants | 19 | 16

5. Secondary Outcome: Number of Frozen Sections Sent for Analysis (of Suspected Parathyroid Tissue).
Description: Number of frozen sections sent for analysis during the procedure to confirm potential parathyroid tissue
Time Frame: Immediate. During total thyroidectomy procedure.
Measure: Mean (Standard Deviation); unit: frozen sections
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
frozen sections | 0.08 (0.4) | 0.1 (0.3)

6. Secondary Outcome: Number of Auto-transplanted Parathyroid Glands
Description: Number of auto-transplanted parathyroid glands if the parathyroid gland was accidentally excised/devascularized.
Time Frame: Immediate. During total thyroidectomy procedure.
Measure: Number; unit: parathyroid glands
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
parathyroid glands | 43 | 39

7. Secondary Outcome: Number of Nights Spent in the Hospital After Total Thyroidectomy
Description: Number of nights spent in the hospital after the surgical procedure. 0 nights, 1 night, >1 night
Time Frame: 0 - 4 nights after total thyroidectomy
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
Participants
  0 Nights | 1 | 4
  1 Night | 77 | 72
  > 1 Night | 2 | 4

8. Secondary Outcome: Number of Inadvertently Resected Parathyroid Glands
Description: Number of inadvertently resected parathyroid glands when parathyroid tissue is found in the resected thyroid specimens.
Time Frame: Intraoperatively or on histology (within 24 hours post operation)
Measure: Mean (Standard Deviation); unit: parathyroid glands
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
Number analyzed (Participants) | 80 | 80
parathyroid glands | 0.09 (0.3) | 0.06 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 2 years and 5 months.
Arm/Group | NIRAF Detection Technology + | NIRAF Detection Technology -
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

LIMITATIONS AND CAVEATS:
The median follow-up time of participants was 5-14 days post-operation. Therefore, we lack long-term follow-up (> 6 months) for the majority of the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT04281875/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT04281875/ICF_001.pdf